CLINICAL TRIAL: NCT00254488
Title: Acute Pharmacotherapy of Late-Life Mania (GERI-BD)
Brief Title: Treatment of Bipolar Mania in Older Adults
Acronym: GERI-BD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U01MH068847 (NIH); U01MH068847 (NIH)
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Results first posted 2018-08-14 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Bipolar Disorder; Mania
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Lithium; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lithium (LI) (Experimental): Participants will receive 9 weeks of treatment with lithium
  Interventions: Drug: Lithium (LI)
- Divalproex (DV) (Experimental): Participants will receive 9 weeks of treatment with divalproex
  Interventions: Drug: Divalproex (DV)

INTERVENTIONS:
Drug: Lithium (LI) — The starting LI dose will be 150 mg in the morning and evening. The dose of medication will be adjusted to achieve plasma LI level ranges between 0.40 and 0.99 mEq/L (target 0.80 to 0.99 mEq/L).
  Other Names: Depakote
  Arms: Lithium (LI)
Drug: Divalproex (DV) — Dosage of DV will be 250 mg in the morning and evening. The dose of medication will be adjusted to achieve plasma DV level ranges between 40 and 99 mcg/mL (target 80 to 99 mcg/ml).
  Other Names: Valproate
  Arms: Divalproex (DV)

SUMMARY:
This study will compare the benefits and side effects of lithium and divalproex in the treatment of older adults with bipolar mania.

DETAILED DESCRIPTION:
This is the first controlled acute treatment study of bipolar disorder in adults 60 years or older with current DSM-IV manic, mixed, or hypomanic episodes. The number of older adults with severe and disabling bipolar disorder is increasing, and information to guide the management of the treatment of the disease is lacking in this population. Guidelines for treatment of younger people with bipolar disorder cannot be used for older people, and there are no safety and efficacy data upon which to base initial treatment decisions for older patients with bipolar mania. Mood stabilizers (lithium and divalproex) are the first-line treatment for bipolar disorder. However, in aged patients physiological changes and comorbid diseases may increase vulnerability to side effects and limit the benefits of the medications.

This double-blind study will compare the benefits and side-effects of 9 weeks of treatment with lithium and divalproex in people with bipolar mania. Participants, who may be treated during inpatient hospitalization or as outpatients, will be randomly assigned to receive either lithium or divalproex. During the first 3 weeks of treatment careful titration of lithium and divalproex will be done to reach dose ranges. All other psychotropic medications will be discontinued. Behavioral interventions and/or lorazepam may be added, if necessary. After the first 3 weeks, if symptoms do not improve, risperidone will be added to be taken everyday with the study medication.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DSM-IV Bipolar Disorder, Type I: current manic, mixed, or hypomanic episodes

Exclusion Criteria:

* Rapid cycling bipolar disorder
* History of substance abuse or dependence within last 3 months
* Diagnosis of schizophrenia or other chronic psychotic conditions
* Acute or unstable medical illness
* Documented intolerance to Lithium, Depakote, Risperidone, or Lorazepam
* Dementia
* Inability to communicate in English

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2005-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Young, MD, Study Chair — Cornell University
Locations (8):
- United States (7):
  - Precise Research Centers, Flowood, Mississippi
  - Weill Cornell Medical College, White Plains, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Result] Al Jurdi RK, Schulberg HC, Greenberg RL, Kunik ME, Gildengers A, Sajatovic M, Mulsant BH, Young RC; GERI-BD Study Group. Characteristics associated with inpatient versus outpatient status in older adults with bipolar disorder. J Geriatr Psychiatry Neurol. 2012 Mar;25(1):62-8. doi: 10.1177/0891988712436684. PMID 22467848
- [Result] Beyer JL, Greenberg RL, Marino P, Bruce ML, Al Jurdi RK, Sajatovic M, Gyulai L, Mulsant BH, Gildengers A, Young RC. Social support in late life mania: GERI-BD. Int J Geriatr Psychiatry. 2014 Oct;29(10):1028-32. doi: 10.1002/gps.4093. Epub 2014 Mar 24. PMID 24664811
- [Result] Sajatovic M, Al Jurdi R, Gildengers A, Greenberg RL, Tenhave T, Bruce ML, Mulsant B, Young RC. Depression symptom ratings in geriatric patients with bipolar mania. Int J Geriatr Psychiatry. 2011 Nov;26(11):1201-8. doi: 10.1002/gps.2664. Epub 2011 Mar 1. PMID 21360754
- [Result] Gildengers AG, Mulsant BH, Al Jurdi RK, Beyer JL, Greenberg RL, Gyulai L, Moberg PJ, Sajatovic M, ten Have T, Young RC; GERI-BD Study Group. The relationship of bipolar disorder lifetime duration and vascular burden to cognition in older adults. Bipolar Disord. 2010 Dec;12(8):851-8. doi: 10.1111/j.1399-5618.2010.00877.x. PMID 21176032
- [Result] Young RC, Schulberg HC, Gildengers AG, Sajatovic M, Mulsant BH, Gyulai L, Beyer J, Marangell L, Kunik M, Ten Have T, Bruce ML, Gur R, Marino P, Evans JD, Reynolds CF 3rd, Alexopoulos GS. Conceptual and methodological issues in designing a randomized, controlled treatment trial for geriatric bipolar disorder: GERI-BD. Bipolar Disord. 2010 Feb;12(1):56-67. doi: 10.1111/j.1399-5618.2009.00779.x. PMID 20148867
- [Derived] Young RC, Mulsant BH, Sajatovic M, Gildengers AG, Gyulai L, Al Jurdi RK, Beyer J, Evans J, Banerjee S, Greenberg R, Marino P, Kunik ME, Chen P, Barrett M, Schulberg HC, Bruce ML, Reynolds CF 3rd, Alexopoulos GS; GERI-BD Study Group. GERI-BD: A Randomized Double-Blind Controlled Trial of Lithium and Divalproex in the Treatment of Mania in Older Patients With Bipolar Disorder. Am J Psychiatry. 2017 Nov 1;174(11):1086-1093. doi: 10.1176/appi.ajp.2017.15050657. Epub 2017 Aug 4. PMID 29088928

RESULTS

PARTICIPANT FLOW:
Groups:
- Lithium: Participants will receive 9 weeks of treatment with lithium
  Lithium (LI): The starting LI dose will be 150 mg in the morning and evening. The dose of medication will be adjusted to achieve plasma LI level ranges between 0.40 and 0.99 mEq/L (target 0.80 to 0.99 mEq/L).
- Divalproex: Participants will receive 9 weeks of treatment with divalproex
  Divalproex (DV): Dosage of DV will be 250 mg in the morning and evening. The dose of medication will be adjusted to achieve plasma DV level ranges between 40 and 99 mcg/mL (target 80 to 99 mcg/ml).
Period: Overall Study
Arm/Group | Lithium | Divalproex
Started | 112 | 112
Completed | 55 | 63
Not Completed | 57 | 49

BASELINE CHARACTERISTICS:
Groups:
- Lithium (LI): Participants will receive 9 weeks of treatment with Lithium. The starting Lithium dose will be 150 mg in the morning and evening.
- Divalproex (DV): Participants will receive 9 weeks of treatment with Divalproex. The starting Divalproex dose will be 250 mg in the morning and evening.
- Total: Total of all reporting groups
Arm/Group | Lithium (LI) | Divalproex (DV) | Total
Number analyzed (Participants) | 112 | 112 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (6.8) | 68.3 (6.1) | 68.0 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 59 | 115
  Male | 56 | 53 | 109
Young Mania Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The Young Mania Rating Scale (YMRS) is an eleven item interviewer-rated instrument. Four items are scored 0-8, the others 0-4. The total score therefore ranges from 0-60, with higher values reflecting greater severity.
  units on a scale | 27.1 (7.4) | 25.5 (6.1) | 26.3 (6.8)
Sedation score [Mean (Standard Deviation); unit: units on a scale] — The Sedation Item score of the UKU (Norwegian for Committee of Clinical Investigations) Side Effect Rating Scale. A higher value indicates greater severity. Range is 0-3 (not present, mild, moderate, or severe).
  units on a scale | .5 (.7) | .5 (.6) | .5 (.65)

OUTCOME MEASURES:

1. Primary Outcome: Sedation Score
Description: The Sedation Item score of the UKU (Norwegian for Committee of Clinical Investigations) Side Effect Rating Scale. A higher value indicates greater severity. Range is 0-3 (not present, mild, moderate, or severe).
Time Frame: Day 4, Day 9, Day 15, and then Weekly from Week 3 to Week 9
Population: The number of participants analyzed over the course of the study decreases due to participants missing a visit or dropping from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lithium (LI) | Divalproex (DV)
Number analyzed (Participants) | 107 | 109
units on a scale
  Day 4 | 0.5 (0.7) | 0.5 (0.7)
  Day 9: number analyzed (Participants) | 105 | 99
  Day 9 | 0.6 (0.7) | 0.6 (0.6)
  Day 15: number analyzed (Participants) | 98 | 95
  Day 15 | 0.4 (0.6) | 0.5 (0.7)
  Week 3: number analyzed (Participants) | 93 | 91
  Week 3 | 0.5 (0.7) | 0.6 (0.7)
  Week 4: number analyzed (Participants) | 75 | 81
  Week 4 | 0.5 (0.7) | 0.5 (0.6)
  Week 5: number analyzed (Participants) | 66 | 78
  Week 5 | 0.5 (0.7) | 0.4 (0.6)
  Week 6: number analyzed (Participants) | 61 | 73
  Week 6 | 0.5 (0.7) | 0.5 (0.6)
  Week 7: number analyzed (Participants) | 60 | 67
  Week 7 | 0.4 (0.6) | 0.4 (0.5)
  Week 8: number analyzed (Participants) | 54 | 63
  Week 8 | 0.4 (0.6) | 0.3 (0.5)
  Week 9: number analyzed (Participants) | 55 | 63
  Week 9 | 0.4 (0.6) | 0.4 (0.6)

2. Primary Outcome: Young Mania Rating Scale (YMRS) Scores
Description: The Young Mania Rating Scale is an eleven item interviewer-rated instrument. Four items are scored 0-8, the others 0-4. The total score therefore ranges from 0-60, with higher values reflecting greater severity.
Time Frame: Day 4, Day 9, Day 15, and then Weekly from Week 3 to Week 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lithium (LI) | Divalproex (DV)
Number analyzed (Participants) | 108 | 109
units on a scale
  Day 4 | 21.4 (9.3) | 19.7 (7.7)
  Day 9: number analyzed (Participants) | 107 | 99
  Day 9 | 19.0 (9.5) | 16.3 (8.1)
  Day 15: number analyzed (Participants) | 96 | 100
  Day 15 | 14.3 (9.3) | 15.2 (8.7)
  Week 3: number analyzed (Participants) | 95 | 92
  Week 3 | 12.1 (8.8) | 13.1 (9.4)
  Week 4: number analyzed (Participants) | 76 | 82
  Week 4 | 9.4 (5.9) | 9.9 (7.1)
  Week 5: number analyzed (Participants) | 68 | 79
  Week 5 | 7.6 (5.8) | 9.8 (7.0)
  Week 6: number analyzed (Participants) | 60 | 73
  Week 6 | 7.2 (5.4) | 8.2 (6.5)
  Week 7: number analyzed (Participants) | 60 | 67
  Week 7 | 6.0 (6.0) | 7.0 (5.9)
  Week 8: number analyzed (Participants) | 54 | 63
  Week 8 | 6.0 (5.4) | 6.7 (5.8)
  Week 9: number analyzed (Participants) | 55 | 63
  Week 9 | 6.3 (6.0) | 6.8 (5.9)

ADVERSE EVENTS:
Time Frame: 9 weeks
Description: Clinicaltrials.gov definitions apply.
Arm/Group | Lithium (LI) | Divalproex (DV)
All-Cause Mortality (participants affected / at risk) | 0/112 | 2/112
Serious Adverse Events (participants affected / at risk) | 24/112 | 22/112
Other Adverse Events (participants affected / at risk) | 69/112 | 70/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium (LI) (N=112) | Divalproex (DV) (N=112)
Psychiatric condition worsening (Psychiatric disorders) | 9 (9) | 11 (12) — Psychiatric Hospitalization due to worsening condition
Elevated liver enzymes (Hepatobiliary disorders) | 0 (0) | 1 (1)
Circulatory condition (Vascular disorders) | 1 (1) | 2 (3)
Chest pain (Cardiac disorders) | 2 (2) | 1 (1)
Suicide (Psychiatric disorders) | 0 (0) | 1 (1) — One completed suicide after study completion
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospitalization for rectal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hospitalization for cellulitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hospitalization for Urinary Tract infection (Infections and infestations) | 0 (0) | 1 (1)
Medical intervention for Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Medical complications due to alcohol abuse (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
numbness (Nervous system disorders) | 1 (1) | 1 (1)
Increased creatine level (Investigations) | 1 (1) | 0 (0)
Unsteady gait with a subsequent fall, increased confusion and tremulousness (General disorders) | 2 (2) | 0 (0)
Edema (General disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Low blood pressure (Vascular disorders) | 1 (1) | 0 (0)
Back surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nausea and vomitting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.89% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium (LI) (N=112) | Divalproex (DV) (N=112)
Elevated glucose (Metabolism and nutrition disorders) | 4 (8) | 0 (0)
Decrease in sodium (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cardiac change (Cardiac disorders) | 6 (6) | 5 (5)
Calcium Deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Change in Thyroid level (Endocrine disorders) | 1 (1) | 0 (0)
Gastrointestinal symptoms (Gastrointestinal disorders) | 24 (33) | 26 (35)
Infection (Infections and infestations) | 4 (6) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 19 (27) | 20 (27)
Accidental injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
weight gain (Investigations) | 13 (14) | 23 (27)
Weight loss (Investigations) | 13 (15) | 6 (6)
Change in pre existing high blood pressure (Investigations) | 0 (0) | 2 (2)
Change in Amylase and Lipase lab values (Investigations) | 6 (8) | 0 (0)
Increased creatine level in lab work (Investigations) | 1 (1) | 0 (0)
Nosebleed (Investigations) | 1 (1) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6)
laboratory finding Increased liver enzymes (Investigations) | 0 (0) | 3 (3)
laboratory findings increased white blood count (Investigations) | 0 (0) | 3 (3)
Worsening psychiatric symptoms (Psychiatric disorders) | 2 (6) | 5 (10)
Elevated blood levels (Renal and urinary disorders) | 0 (0) | 4 (4)
Urinary dysfunction (Renal and urinary disorders) | 6 (6) | 3 (3)
Sexual dysfunction (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 6 (6)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (8)
Hypertension (Vascular disorders) | 3 (5) | 4 (7)
Vision disturbance (Eye disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 7 (10) | 2 (4)
Sedation (Nervous system disorders) | 7 (7) | 3 (5)
Decreased need for sleep (Nervous system disorders) | 1 (1) | 1 (1)
Memory Change (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 3 (4)
Dizziness (Nervous system disorders) | 3 (4) | 1 (2)
Restlessness (Nervous system disorders) | 2 (2) | 1 (1)
Sinus tension (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes